CLINICAL TRIAL: NCT04141618
Title: Dr. Pao-Lin Kuo (Department of Obstetrics and Gynecology)
Brief Title: The Role of NLRP Gene Family (NLRP1~14) in Recurrent Miscarriage and Infertility
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BR-100-006
Record Dates: First submitted 2014-04-07; First posted 2019-10-28 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2019-10

CONDITIONS: Miscarriage, Recurrent; Infertility
Keywords: recurrent miscarriage; infertility
MeSH Terms: conditions — Abortion, Habitual; Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA extracted from peripheral blood.

SUMMARY:
Development of mole was not associated with segregation of mutated NLRP7 allele in the haploid oocyte. We hypothesize NLRP7 is a maternal factor involved in regulating early embryo development or embryo-uterine interaction. In the proposed study, we seek to identify novel genetic variants and mutations of NLRP7 in women who experienced RM/HM. Genetic association study and haplotype analysis are performed to test assocation between NLRP7 gene and female reproductive performance. Immunohistochemical staining, RT-PCR, and Western blot analysis are used to investigate expression pattern of NLRP7 in endometrium and placenta. Two approaches are used to characterize functional significance of genetic variants/mutations. The first approach will be based on mutagenesis and the second approach will be based on induced pluripotent stem cells (iPSCs). Results obtained from the proposed study will provide novel insight into mechanism of embryo development and implantation.

DETAILED DESCRIPTION:
Recurrent miscarriage (RM), defined as at least two consecutive fetal death or spontaneous abortions before the 20th week gestational age, occurred in about 1% to 5% couples. The causes of RM include uterine factors, endocrine factors, thromobophilic factors, immunologic factors and genetic factors. The hydatidiform mole (HM) can be divided into two separate syndromes: complete mole (CHM) and partial mole (PHM). In the West, CHMs occur in approximately 1 in every 1500 pregnancies. The incidence is higher in Latin America, Southeast Asia and the Middle East. The cause of RM and HM are not known for the vast majority of cases. The NLRP (Nucleotide-binding oligomerization domain, Leucine rich Repeat and Pyrin domain containing) family, also referred to as NALP family, is well known for its roles in apoptosis and inflammation. Expression studies showed that twelve of the fourteen members of NLRP family express differentially in human oocytes and preimplantation embryonic cells, especially NLRP7, indicating important role of NLRP family in female reproduction. Since 2006, mutations of NLRP7 have been found in women with repeated occurrence of molar pregnancy, repeated stillbirth or early spontaneous abortion. In women who experienced RM/HM, we also found some novel mutations/genetic variants of NLRP7. Taken together, these finding suggest RM and HM may share the same genetic etiology in some cases. In addition, NLRP7 is a strong candidate gene for RM/HM. A recent report showed chaotic cleavage abnormalities of embryos in patients with NLRP7 variants.

ELIGIBILITY:
Inclusion Criteria:

Recurrent abortions and infertility treatments but combined with repetitive (more than two consecutive) implantation failure couples, rather than general infertility couples.

Exclusion Criteria:

Women who do not have recurrent miscarriage and infertility problems.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Assuming that there are 300 cases and 300 controls enrolled, the underlying disease model is recessive, the disease prevalence is approximately 3% and the disease allele frequency is about 5%, this study has more than 80% power for detecting the SNP with an allele frequency greater than 10% and an allelic odds ratio greater than 1.4. We assumed that the SNP is either the causal gene or in LD with the causal allele and power was calculated without multiple testing corrections.
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2011-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
pregnancy outcome | 1 month at the end of pregnancy
  Pregnancy and delivery of a normal baby is defined as normal outcome

SECONDARY OUTCOMES:
spontaneous abortion | abortion before 12 weeks of gestation
  fail to maintain pregnancy beyond 12 weeks

OTHER OUTCOMES:
intrauterine fetal death | fetal death after 12 weeks of gestation
  pregnancy beyond 12 weeks followed by death of the fetus

CONTACTS AND LOCATIONS:
Overall Officials: Pao-Lin Kuo, MD, Principal Investigator — Department of Obstetrics and Gynecology, National Cheng Kung University Hospital
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan